CLINICAL TRIAL: NCT02882815
Title: Post Market Clinical Follow-up Study of IrisFITTM PFO (Patent Foramen Ovale)
Brief Title: Post Market Clinical Follow-up Study of IrisFITTM PFO (Patent Foramen Ovale) Occluder
Acronym: PFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFO-01
Record Dates: First submitted 2016-08-03; First posted 2016-08-30 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Patent Foramen Ovale
Keywords: IrisFIT PFO
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IrisFIT PFO Occluder (Other): Participating patients will have their PFO closed using the IrisFITTM PFO Occluder device.The patients will undergo a clinical examination, electrocardiogram (ECG), clinical laboratory assessment and transthoracic echocardiography (TTE). All periprocedural procedures will be performed according to site´s standard of care.. The efficacy and safety of the devices will be assessed by ECGs, vital signs, physical examination and TTE, which will be done at 1day, at 1month and at 6 months post procedure. Safety will also be assessed at 12 months by telephone visit.
  Interventions: Device: IrisFIT PFO Occluder

INTERVENTIONS:
Device: IrisFIT PFO Occluder

SUMMARY:
The purpose of the study is to collect more data about performance and safety of the device called "IrisFITTM PFO occluder". This data will be used to help more patients who will accept treatment with this device in the future.

Patients will undergo routine examination, procedure and follow-up. Related data will be collected and kept in a way that patient info is well protected.

DETAILED DESCRIPTION:
This is a Post Market Clinical Follow-up study. Informed consent will be obtained from the patient or from a legally authorized representative of the patient at screening. The patients will be screened (pre-procedure) to determine eligibility for the study. At screening, patients will be assessed for study eligibility by the inclusion/exclusion criteria through their medical history, demographics and transthoracic echocardiography (TTE). Participating patients will have their PFO closed using the IrisFITTM PFO Occluder device. The patients will undergo a clinical examination, electrocardiogram (ECG), clinical laboratory assessment and transthoracic echocardiography (TTE). All periprocedural procedures will be performed according to site´s standard of care.. The efficacy and safety of the devices will be assessed by ECGs, vital signs, physical examination and TTE, which will be done at 1day, at 1month and at 6 months post procedure. Safety will also be assessed at 12 months by telephone visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are according to current international or local guidelines (and future revisions) and per physician discretion scheduled for interventional treatment of PFO.
* Patients who are willing and capable of providing informed consent and participating in all testing/or follow procedure associated with this study.
* Patients who are eligible for treatment with IrisFIT PFO occluder device. (Per physician discretion and device IFU).

Exclusion Criteria:

* PFO tunnel length <1 mm
* Women of childbearing potential who are or plan to become pregnant during the time of the study (method of assessment upon physician's discretion)
* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Adverse device effects during the procedure up to the point of implanting the study device in the PFO, and during completion of the procedure | during completion of the procedure
  Adverse device effects during the procedure up to the point of implanting the study device in the PFO, and during completion of the procedure
Device related adverse event up to 1 month follow-up | 1 month post procedure
  Device related adverse event up to 1 month follow-up
Device related adverse event up to 12 month follow-up | 12 month post procedure
  Device related adverse event up to 12 month follow-up
Rate of accurate device placement | 6 month post procedure
  Rate of accurate device placement
Incidence of device migration/malfunction | 6 month post procedure
  Incidence of device migration/malfunction
Successful closure/procedure rate: Proper position of the occluder by imaging, with trivial to small or without residual shunt, 6 month after procedure). | 6 month post procedure
  Successful closure/procedure rate: Proper position of the occluder by imaging, with trivial to small or without residual shunt, 6 month after procedure).

CONTACTS AND LOCATIONS:
Overall Officials: HORST SIEVERT, Principal Investigator — CARDIOVÄSCULARES CENTRUM FRANKFURT GERMANY
Locations (3):
- Germany (2):
  - Cardio Vasculäres Centrum Frankfurt, Frankfurt
  - Helmut-G.-Walther-Klinikum, Lichtenfels
- Mater Misericordiae University Hospital, Dublin, Ireland